CLINICAL TRIAL: NCT07162103
Title: Investigating the Effects of Group Mandala Art Therapy on Psychological Well-Being and Loneliness Levels in the Elderly
Brief Title: Group Mandala Art Therapy for Well-Being and Loneliness in the Elderly (GEMEL-WB:RCT)
Acronym: GEMEL-WB:RCT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Suleyman Demirel University (Other)
Responsible Party: Principal Investigator, Sema Soysal, Lecturer, Suleyman Demirel University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 24-04-2025/ 95 /11
Record Dates: First submitted 2025-08-28; First posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Elderly Individuals Aged 60 Years or Older
Keywords: Elderly; Psychological well-being; Loneliness; Mandala
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Who Masked: Participant
Masking Description: In this study, researcher blinding will not be performed because the researchers who implemented the intervention and evaluated the data are the project managers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Twelve sessions of group mandala art therapy (GMART)will be applied to the intervention group once a week, and a pretest will be taken in the first session and a posttest will be taken after the 12th week using the "Loneliness Scale for the Elderly" and the "Psychological Well-Being Scale for the Elderly".
  Interventions: Other: GMART
- Control Group (No Intervention): The control group will not receive any intervention, and pretest and posttest data will be collected after the first and 12 weeks using the "Loneliness Scale for the Elderly" and "Psychological Well-Being Scale for the Elderly."

INTERVENTIONS:
Other: GMART — Group Mandala Art Therapy
  Arms: Intervention Group

SUMMARY:
The research is being conducted at an elderly day care center between June 12 and August 31, 2025, as a single-blind randomized controlled experimental study using a pre-test, post-test design. Prior to the research, approval was obtained from the scale owners, the participants, the ethics committee, and the institution's implementation permit. The research population consists of 300 individuals registered at the institution. The study sample will consist of 58 individuals (intervention-29 and control-29) who met the inclusion criteria, were selected using the block randomization method, and provided informed consent. The control group will not receive any intervention, and a pre-test will be administered on the first day, and a post-test will be administered on the day the intervention for the experimental group concluded (Week 12). The intervention group will receive 12 sessions of group mandala art therapy once a week, with a pre-test on the first day and a post-test in the last session (Week 12) following the intervention. Data will be collected using the Personal Information Form (PIF) (Appendix 1), Standardized Mini Mental Test, Psychological Well-Being Scale for the Elderly (YPİOÖ), and Loneliness Scale for the Elderly. Data will be analyzed using the SPSS (Statistical Program for Social Sciences) statistical analysis package program, with statistical significance considered at p <0.05.

DETAILED DESCRIPTION:
The problems associated with aging and the increasing elderly population have led to an increase in the healthcare and rehabilitation needs of older individuals, and the psychosocial health of older individuals has become a global public health concern. Elderly individuals living in nursing homes, in particular, need health promotion activities that will improve their emotional well-being, cognitive status, and physical condition, or reduce problematic behaviors. In this context, art therapy, a supportive method aligned with the biopsychosocial approach, is recommended for interventions aimed at protecting and improving the mental health of older individuals. Art therapy, included in the Nursing Intervention Classification, is a supportive method that helps individuals express themselves, acquire coping skills, develop interpersonal skills, increase resilience, resolve conflicts and problems, manage their behaviors, reduce stress, increase self-esteem and self-confidence, and gain insight using art as a tool, all contributing to psychological well-being. Some studies have emphasized the impact of art-related activities on the health of older individuals. According to the literature, utilizing art in individual or group work with older individuals improves their physical and psychosocial health, reduces functional impairments, increases life satisfaction and quality, and enhances self-confidence. It is suggested that mandala creation, a frequently used technique in art therapy, not only provides insight into certain dynamics underlying an individual's subconscious, such as anxiety, fear, and internal conflicts, but also positively impacts the individual's "healing" process. Mandala is considered by art psychotherapists as a psychotherapy technique that provides psychological support and healing.

Maintaining active social relationships among older individuals is important for preventing feelings of loneliness, a symptom of a lack of social relationships, and for increasing psychological well-being. Social relationships can be maintained through close connections with the environment or through hobbies and recreational activities. The purpose of this study is to examine the effects of mandala art therapy group practices on the levels of loneliness and psychological well-being of older individuals living in nursing homes. Consequently, since its inception, nursing has prioritized the holistic healing and recovery of individuals under its care and responsibility, grounded in an existential-humanistic understanding. Since Florence Nightingale, considered the founder of environmental interaction theory and modern nursing, therapeutic management of an individual's environment and setting has held a prominent place among nurses' roles and responsibilities. In this sense, creating a healing/therapeutic environment is a fundamental component of nursing care. In this context, nurses must provide a healing environment enriched with activities to maintain and support the well-being of older individuals, their sense of meaning and purpose in life. Therefore, in the face of a rapidly aging population, encouraging the use of evidence-based interventions to enhance or maintain the well-being of older individuals is crucial. No studies have been found in the literature examining the levels of loneliness and psychological well-being in older individuals using single mandala art therapy. This study has several strengths, including the inclusion of intervention and non-intervention groups, the consistency of the frequency and number of group sessions and materials with the literature, and the examination of comprehensive variables within the life cycle of older adults, such as loneliness and psychological well-being. It is also believed to make significant contributions to the fields of geriatric psychology and art therapy.

In line with the purpose of the study, the hypotheses are as follows:

Hypothesis 1 (H1): Elderly individuals who received group mandala art therapy will have higher post-intervention well-being levels than the control group.

Hypothesis 2 (H1): Elderly individuals who received group mandala art therapy will have lower post-intervention loneliness levels than the control group.

Hypothesis 3 (H1): There is a negative relationship between the well-being and loneliness levels of elderly individuals who received and did not receive group mandala art therapy.

Research Conduct A preliminary study will be conducted with one participant to determine the effectiveness and duration of the measurement tools and group mandala art therapy sessions. The study will be conducted in an elderly daycare center as a single-blind randomized controlled experimental study with a pretest-posttest design. Participants will be provided with an Informed Consent Form and surveys at the beginning of the first session. All participants will complete the surveys at the pretest level and will then be randomized into one of two groups. The control group will not receive any intervention; a posttest will be administered three months after the initial measurements. The control group will also receive the intervention after the research period is concluded. The experimental group will receive the intervention; a posttest will be administered three months after the initial measurements. The study, which will be conducted face-to-face, is planned to consist of twelve (12) sessions, each 90-minute session, once a week for the experimental group. No intervention will be administered to the control group.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer to participate in the study
* No special conditions that would cause cognitive difficulties (auditory or visual impairments, etc.)
* Standardized Mini Mental State Examination (SMMT) score: 23-30 points (no cognitive impairment or mild cognitive impairment)

Exclusion Criteria:

* Presence of a mental or physical disability that prevents communication and attendance at sessions (inability to speak, severe dementia, etc.) Study Exclusion Criteria Indicated desire to withdraw from the study
* Failure to attend a maximum of 3 sessions
* Withdrawal from the institution

Ages: 60 Years to 84 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2025-09-03 (Estimated); Primary Completion 2025-11-05 (Estimated); Study Completion 2025-11-12 (Estimated)

PRIMARY OUTCOMES:
"Loneliness Scale for the Elderly" | Measurements will be made before the first session when the research begins and 12 weeks after the beginning.
  The extent to which a person experiences the situation described in each statement on the scale is determined using a 3-point Likert-type scale. The scale is rated as follows: 0 = yes, 1 = maybe, 2 = no. Responses are made by selecting the rating statement that best describes the individual. Five of the scale items are coded linearly, and six are reverse-coded. The items belonging to the social loneliness sub-dimension (1, 4, 7, 8, and 11), which contain positive expressions, are scored as 0 = yes, 1 = maybe, 2 = no; the items belonging to the emotional loneliness sub-dimension (2, 3, 5, 6, 9, and 10), which contain negative expressions, are scored as 2 = yes, 1 = maybe, 0 = no. The lowest possible score on the scale is 0, and the highest is 22. Total loneliness can be divided into four levels: Level 1: Not lonely/does not feel lonely (scores 0-4); Level 2: Acceptable loneliness (score 5-14); Level 3: Very lonely (score 15-18); Level 4: Very intense loneliness (score 19-22)

SECONDARY OUTCOMES:
"Psychological Well-Being Scale for the Elderly" | Measurements will be made before the first session when the research begins and 12 weeks after the beginning.
  It is a self-reported, 5-point Likert-type scale (1 = completely disagree - 5 = completely agree) that measures psychological well-being in older adults. There is no cut-off score for well-being in older adults based on the scale's scoring. Increasing scores indicate increasing well-being. The minimum score on the scale is 15, and the maximum score is 75.

IPD SHARING:
Plan to Share IPD: Undecided